CLINICAL TRIAL: NCT05026164
Title: A Randomized, Double-Blind, Placebo-Controlled, Repeated-Dose Study to Assess the Safety, Tolerability, and Effects of CHI-202 to Support Recovery From Physical Activity
Brief Title: Study to Assess the Safety, Tolerability, and Effects of CHI-202 to Support Recovery From Physical Activity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canopy Growth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 710US-1311
Record Dates: First submitted 2021-07-26; First posted 2021-08-30 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Delayed Onset Muscle Soreness (DOMS)

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): CHI-202. Participants will drink one 7.0g CHI-202 powder sachet mixed into 16oz of water twice daily.
  Interventions: Dietary Supplement: CHI-202
- Placebo (Placebo Comparator): CHI-101. Participants will drink one 7.0g CHI-101 powder sachet mixed into 16oz of water twice daily.
  Interventions: Dietary Supplement: CHI-101

INTERVENTIONS:
Dietary Supplement: CHI-202 — Blend of cannabinoids & other ingredients
  Arms: Active
Dietary Supplement: CHI-101 — Placebo
  Arms: Placebo

SUMMARY:
The study is designed as a proof of concept, single-center, randomized, double-blind, placebo controlled study to assess the safety and efficacy of CHI-202 (cannabinoids and other ingredients) compared to placebo in the treatment of Delayed Onset Muscle Soreness (DOMS).

DETAILED DESCRIPTION:
The study is designed as a proof of concept, single-center, randomized, double-blind, placebo controlled study to assess the safety and efficacy of CHI-202 (cannabinoids and other ingredients) compared to placebo in the treatment of Delayed Onset Muscle Soreness (DOMS). Healthy adults ages 18-65 years who are exercise-trained (self-report exercising at least 3 times per week for at least 30 minutes per session for the past year) will be recruited from existing panels of participants from past studies, local advertisements, and social media targeted advertisements. Those who meet the inclusion/exclusion criteria will be enrolled into the study, scheduled for the Exercise Visit (Study Visit 1; Day 0) within 2 weeks of screening, and randomized to active vs. placebo IP condition in a 1:1 ratio. One repetition maximum (1RM) method, the maximum amount of weight one can lift in a single repetition for a given exercise, will be used in order to induce DOMS. Following the completion of the Exercise Visit, participants will be scheduled for 3 follow-up visits that will occur 1, 2, and 3 days post-Exercise Visit. Participants will consume 7 scheduled doses of the study IP to which they have been randomly assigned (i.e., active or placebo) with instruction to consume the study IP prior to the exercise at Study Visit 1, at 8PM (±1 hour) that night, and then at 8AM and 8PM (±1 hour) every day until their final study visit. The last dose will occur at 8AM (±1 hour) on Day 4, i.e., immediately prior to Study Visit 4.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy adult aged 18-65 years, inclusive, at the time of screening.
2. Is exercise-trained, i.e., self-reports exercising at least 3 times per week for at least 30 minutes per session for the past year.
3. Has a body mass index between 18 and 35 kg/m2 (inclusive).
4. Is judged by the Investigator to be in generally good health at screening based on participants' self-reported medical history.
5. Must be adequately informed of the nature and risks of the study and give written informed consent prior to screening.

Exclusion Criteria:

1. Women who are pregnant, lactating, breastfeeding, or planning a pregnancy.
2. Women of childbearing potential, or men who are sexually active with a woman of childbearing potential, who are unwilling or unable to use an acceptable method of contraception (abstinence or the use of a highly effective method of contraception, including hormonal contraception, diaphragm, cervical cap, vaginal sponge, condom, vasectomy, or intrauterine device) from at least 21 days prior to the first dose of study medication until 28 days after the last dose of study medication.
3. Has a history of epilepsy, hepatitis, clinically significant hepatic or renal impairment, or human immunodeficiency virus.
4. Changes in the use of a prescription, over-the-counter (OTC), systemic or topical drug(s), herbal supplement(s), or vitamin(s) for the month prior to the Exercise Visit.
5. Has any clinically significant condition or abnormal finding at screening that would, in the opinion of the Investigator, preclude study participation or interfere with the evaluation of the study IP.
6. Has a history of a known significant allergic condition, significant drug-related hypersensitivity, or allergic reaction to any compound or chemical class related to cannabis, including phytocannabinoids and cannabinoid analogues, or excipients utilized within the IP (e.g., coconut; coconut oil; medium-chain triglycerides).
7. Has musculoskeletal issues that might impede performing maximal elbow flexion exercises.
8. Has taken a medication with likely CBD-interactions, including warfarin, clobazam, valproic acid, phenobarbital, mTOR inhibitors, oral tacrolimus, and St. John's Wort within 30 days of the Exercise Visit or during the study.
9. Has taken grapefruit products and/or Seville oranges within the 7 days prior to dosing with study IP.
10. Has used cannabis, synthetic cannabinoid or cannabinoid analogues (e.g., dronabinol, nabilone), hemp products, synthetic cannabinoid receptor agonists (e.g., spice, K2), or any CBD- or THC-containing product (e.g., Sativex, Epidiolex) within 4 weeks of the Exercise Visit or during the study.
11. Has a history or current diagnosis of a significant psychiatric disorder that would, in the opinion of the Investigator, affect the subject's ability to comply with the study requirements.
12. Endorses current suicidal intent.
13. Has participated in any investigational product or device study within 30 days prior to the Screening Visit, or is scheduled to participate in another investigational product or device study during the course of this study.
14. Demonstrates behavior indicating unreliability or inability to comply with the requirements of the protocol.
15. Has a positive result on urine drug screen for cocaine, amphetamine, methamphetamine, THC, and opiates at the first study visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in blood pressure (mmHg) [Safety and Tolerability] | Day 2
  Blood pressure is measure by the combination of systolic and diastolic measurements
Changes from baseline in blood pressure (mmHg) [Safety and Tolerability] | Day 3
  Blood pressure is measure by the combination of systolic and diastolic measurements
Changes from baseline in blood pressure (mmHg) [Safety and Tolerability] | Day 4
  Blood pressure is measure by the combination of systolic and diastolic measurements
Changes from baseline in respiratory rate (breaths per minute) [Safety and Tolerability] | Day 2
  Respiratory rate will be measured as breaths per minute
Changes from baseline in respiratory rate (breaths per minute) [Safety and Tolerability] | Day 3
  Respiratory rate will be measured as breaths per minute
Changes from baseline in respiratory rate (breaths per minute) [Safety and Tolerability] | Day 4
  Respiratory rate will be measured as breaths per minute
Changes from baseline in heart rate (beats per minute) [Safety and Tolerability] | Day 2
  Heart rate will be measured as heart beats per minute
Changes from baseline in heart rate (beats per minute) [Safety and Tolerability] | Day 3
  Heart rate will be measured as heart beats per minute
Changes from baseline in heart rate (beats per minute) [Safety and Tolerability] | Day 4
  Heart rate will be measured as heart beats per minute
Total number of Adverse Events [Safety and Tolerability] | Through study completion (Day 4)
  Safety and tolerability will be assessed through Adverse Events and Serious Adverse Events
Total number of participants with Adverse Events [Safety and Tolerability] | Through study completion (Day 4)
  Safety and tolerability will be assessed through Adverse Events and Serious Adverse Events
Compliance with IP consumption (total # of self-reported doses consumed/maximum of 7 total possible doses consumed) [Safety and Tolerability] | Through study completion (Day 4)
  Safety and tolerability will be assessed through Compliance with IP consumption (total # of self-reported doses consumed/maximum of 7 total possible doses consumed)

SECONDARY OUTCOMES:
Average soreness or discomfort intensity using the 11-point (0-10) NRS | Day 1 - post DOMS intervention
  Self-reported average soreness or discomfort intensity using 11-point (0-10) NRS where 10 is most soreness/discomfort intensity
Average soreness or discomfort intensity over the last 24 hours using the 11-point (0-10) NRS | Day 2
  Self-reported average soreness or discomfort intensity over the last 24 hours using 11-point (0-10) NRS where 10 is most soreness/discomfort intensity
Average soreness or discomfort intensity over the last 24 hours using the 11-point (0-10) NRS | Day 3
  Self-reported average soreness or discomfort intensity over the last 24 hours using 11-point (0-10) NRS where 10 is most soreness/discomfort intensity
Average soreness or discomfort intensity over the last 24 hours using the 11-point (0-10) NRS | Day 4
  Self-reported average soreness or discomfort intensity over the last 24 hours using 11-point (0-10) NRS where 10 is most soreness/discomfort intensity
Worst soreness or discomfort intensity using the 11-point (0-10) NRS | Day 1 - post DOMS intervention
  Self-reported worst soreness or discomfort intensity using the 11-point (0-10) NRS where 10 is most soreness/discomfort intensity
Worst soreness or discomfort intensity over the last 24 hours using the 11-point (0-10) NRS | Day 2
  Self-reported worst soreness or discomfort intensity over the last 24 hours using the 11-point (0-10) NRS where 10 is most soreness/discomfort intensity
Worst soreness or discomfort intensity over the last 24 hours using the 11-point (0-10) NRS | Day 3
  Self-reported worst soreness or discomfort intensity over the last 24 hours using the 11-point (0-10) NRS where 10 is most soreness/discomfort intensity
Worst soreness or discomfort intensity over the last 24 hours using the 11-point (0-10) NRS | Day 4
  Self-reported worst soreness or discomfort intensity over the last 24 hours using the 11-point (0-10) NRS where 10 is most soreness/discomfort intensity
Average stiffness intensity using the 11-point (0-10) NRS | Day 1 - post DOMS intervention
  Self-reported average stiffness intensity using the 11-point (0-10) NRS where 10 is most stiffness intensity
Average stiffness intensity over the last 24 hours using the 11-point (0-10) NRS | Day 2
  Self-reported average stiffness intensity over the last 24 hours using the 11-point (0-10) NRS where 10 is most stiffness intensity
Average stiffness intensity over the last 24 hours using the 11-point (0-10) NRS | Day 3
  Self-reported average stiffness intensity over the last 24 hours using the 11-point (0-10) NRS where 10 is most stiffness intensity
Average stiffness intensity over the last 24 hours using the 11-point (0-10) NRS | Day 4
  Self-reported average stiffness intensity over the last 24 hours using the 11-point (0-10) NRS where 10 is most stiffness intensity
Worst stiffness intensity using the 11-point (0-10) NRS | Day 1 - post DOMS intervention
  Self-reported worst stiffness intensity using the 11-point (0-10) NRS where 10 is most stiffness intensity
Worst stiffness intensity over the last 24 hours using the 11-point (0-10) NRS | Day 2
  Self-reported worst stiffness intensity over the last 24 hours using the 11-point (0-10) NRS where 10 is most stiffness intensity
Worst stiffness intensity over the last 24 hours using the 11-point (0-10) NRS | Day 3
  Self-reported worst stiffness intensity over the last 24 hours using the 11-point (0-10) NRS where 10 is most stiffness intensity
Worst stiffness intensity over the last 24 hours using the 11-point (0-10) NRS | Day 4
  Self-reported worst stiffness intensity over the last 24 hours using the 11-point (0-10) NRS where 10 is most stiffness intensity
Interference of soreness, discomfort, or stiffness after exercise on the ability to perform daily activities at home or at work over the last 24 hours using the 11-point (0-10) NRS | Day 2
  Self-reported interference of soreness, discomfort, or stiffness after exercise on the ability to perform daily activities at home or at work over the last 24 hours using the 11-point (0-10) NRS where 10 is most interference
Interference of soreness, discomfort, or stiffness after exercise on the ability to perform daily activities at home or at work over the last 24 hours using the 11-point (0-10) NRS | Day 3
  Self-reported interference of soreness, discomfort, or stiffness after exercise on the ability to perform daily activities at home or at work over the last 24 hours using the 11-point (0-10) NRS where 10 is most interference
Interference of soreness, discomfort, or stiffness after exercise on the ability to perform daily activities at home or at work over the last 24 hours using the 11-point (0-10) NRS | Day 4
  Self-reported interference of soreness, discomfort, or stiffness after exercise on the ability to perform daily activities at home or at work over the last 24 hours using the 11-point (0-10) NRS where 10 is most interference
Interference of soreness, discomfort, or stiffness after exercise on the ability to participate in physical activities over the last 24 hours using the 11-point (0-10) NRS | Day 2
  Self-reported interference of soreness, discomfort, or stiffness after exercise on the ability to participate in physical activities over the last 24 hours using the 11-point (0-10) NRS where 10 is most interference
Interference of soreness, discomfort, or stiffness after exercise on the ability to participate in physical activities over the last 24 hours using the 11-point (0-10) NRS | Day 3
  Self-reported interference of soreness, discomfort, or stiffness after exercise on the ability to participate in physical activities over the last 24 hours using the 11-point (0-10) NRS where 10 is most interference
Interference of soreness, discomfort, or stiffness after exercise on the ability to participate in physical activities over the last 24 hours using the 11-point (0-10) NRS | Day 4
  Self-reported interference of soreness, discomfort, or stiffness after exercise on the ability to participate in physical activities over the last 24 hours using the 11-point (0-10) NRS where 10 is most interference
Self-reported sleep quality using the 11-point (0-10) NRS | Day 2
  Self-reported sleep quality using the 11-point (0-10) NRS where 10 is best sleep quality
Self-reported sleep quality using the 11-point (0-10) NRS | Day 3
  Self-reported sleep quality using the 11-point (0-10) NRS where 10 is best sleep quality
Self-reported sleep quality using the 11-point (0-10) NRS | Day 4
  Self-reported sleep quality using the 11-point (0-10) NRS where 10 is best sleep quality
Self-reported sleep duration via a sleep diary | Day 2
  Self-reported sleep duration measured in minutes via a sleep diary
Self-reported latency to sleep onset via a sleep diary | Day 2
  Self-reported latency to sleep onset measured in minutes via a sleep diary
Self-reported sleep continuity via a sleep diary | Day 2
  Self-reported sleep continuity measured in minutes via a sleep diary
Self-reported alertness upon waking via a sleep diary | Day 2
  Self-reported alertness upon waking via a sleep diary. Alertness is measure on a scale of 1 to 3 where 1 is Alert, 2 is Alert but a little tired and 3 is Sleepy
Self-reported sleep duration via a sleep diary | Day 3
  Self-reported sleep duration measured in minutes via a sleep diary
Self-reported latency to sleep onset via a sleep diary | Day 3
  Self-reported latency to sleep onset measured in minutes via a sleep diary
Self-reported sleep continuity via a sleep diary | Day 3
  Self-reported sleep continuity measured in minutes via a sleep diary
Self-reported alertness upon waking via a sleep diary | Day 3
  Self-reported alertness upon waking via a sleep diary. Alertness is measure on a scale of 1 to 3 where 1 is Alert, 2 is Alert but a little tired and 3 is Sleepy
Self-reported sleep duration via a sleep diary | Day 4
  Self-reported sleep duration measured in minutes via a sleep diary
Self-reported latency to sleep onset via a sleep diary | Day 4
  Self-reported latency to sleep onset measured in minutes via a sleep diary
Self-reported sleep continuity via a sleep diary | Day 4
  Self-reported sleep continuity measured in minutes via a sleep diary
Self-reported alertness upon waking via a sleep diary | Day 4
  Self-reported alertness upon waking via a sleep diary. Alertness is measure on a scale of 1 to 3 where 1 is Alert, 2 is Alert but a little tired and 3 is Sleepy
Pressure threshold | Day 1 - post DOMS intervention
  Pressure threshold measured with a 25-lb algometer
Pressure threshold | Day 2
  Pressure threshold measured with a 25-lb algometer
Pressure threshold | Day 3
  Pressure threshold measured with a 25-lb algometer
Pressure threshold | Day 4
  Pressure threshold measured with a 25-lb algometer
Relaxed elbow angle | Day 1 - post DOMS intervention
  Relaxed elbow angle measured with a goniometer in degrees
Active range of motion | Day 1 - post DOMS intervention
  Active range of motion measured with a goniometer in degrees
Passive range of motion | Day 1 - post DOMS intervention
  Passive range of motion measured with a goniometer in degrees
Relaxed elbow angle | Day 2
  Relaxed elbow angle measured with a goniometer in degrees
Active range of motion | Day 2
  Active range of motion measured with a goniometer in degrees
Passive range of motion | Day 2
  Passive range of motion measured with a goniometer in degrees
Relaxed elbow angle | Day 3
  Relaxed elbow angle measured with a goniometer in degrees
Active range of motion | Day 3
  Active range of motion measured with a goniometer in degrees
Passive range of motion | Day 3
  Passive range of motion measured with a goniometer in degrees
Relaxed elbow angle | Day 4
  Relaxed elbow angle measured with a goniometer in degrees
Active range of motion | Day 4
  Active range of motion measured with a goniometer in degrees
Passive range of motion | Day 4
  Passive range of motion measured with a goniometer in degrees
Muscle circumference | Day 1 - post DOMS intervention
  Muscle circumference
Muscle circumference | Day 2
  Muscle circumference
Muscle circumference | Day 3
  Muscle circumference
Muscle circumference | Day 4
  Muscle circumference
Mood using the Profile of Mood States | Day 1 - post DOMS intervention
  Mood using the Profile of Mood States
Mood using the Profile of Mood States | Day 2
  Mood using the Profile of Mood States
Mood using the Profile of Mood States | Day 3
  Mood using the Profile of Mood States
Mood using the Profile of Mood States | Day 4
  Mood using the Profile of Mood States

CONTACTS AND LOCATIONS:
Overall Officials: Erica Peters, PhD, Study Director — Canopy Growth Corporation
Locations (1):
- International Society for Sports Nutrition, Boca Raton, Florida, United States